CLINICAL TRIAL: NCT02306772
Title: An Open Label, Single-site Pharmaco-Scintigraphic Study in Healthy Subjects With Radio-labelled TP05-tablets (Mesalazine) to Evaluate the Gastrointestinal Transit and Release Profiles of Two Different Formulations.
Brief Title: TP0501 - Pharmaco-Scintigraphic-Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TP0501
Record Dates: First submitted 2014-10-15; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental): TP05 Coating A
  Interventions: Drug: TP05 Coating A
- Formulation B (Experimental): TP05 Coating B
  Interventions: Drug: TP05 Coating B

INTERVENTIONS:
Drug: TP05 Coating A — One radio-labelled tablet given to subjects
  Other Names: Mesalazine
  Arms: Formulation A
Drug: TP05 Coating B — One radio-labelled tablet given to subjects
  Other Names: Mesalazine
  Arms: Formulation B

SUMMARY:
This is a Phase I, open-label, single-site trial to evaluate the drug release, using Scintigraphic images and mesalazine plasma levels (PK) in healthy subjects. Overall, nine [9] subjects per prototype coating (a total of 18) will be evaluated. Eligible subjects will be assigned in a 1:1 ratio to receive radio-labelled TP05; the first 9 subjects will receive formulation B and the second 9 subjects will receive formulation A. The subjects will be treated once with the radio-labelled study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male or non-pregnant, non-lactating females, between 18 and 55 years old. Females of child bearing potential must have a negative serum pregnancy test prior to the intake of study drug, and must use a hormonal (oral, implantable or injectable) or a double barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. Ability of subject to participate fully in all aspects of this clinical trial.
3. Voluntarily signed informed consent must be obtained and documented.

Exclusion Criteria:

1. Participating in a clinical study involving investigational drugs or dosage forms within the previous 2 months.
2. History of alcohol or drug abuse.
3. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-ray but excluding background radiation, exceeds 5 mSV in the last 12 months or 10 mSv in the last 5 years. No subject whose occupational exposure is monitored will participate in the study.
4. Any nuclear medicine procedure prior to study day 1 that might interfere with the scintigraphic images that are acquired.
5. Clinically significant abnormal biochemistry, haematology or urine analyses:

   * White blood count < 3 x 109/L and > 8 x 109/L
   * Lymphocyte count < 0.85 x 109/L
   * Haemoglobin < 110 g/L
   * Platelet count < 125 x 109/L or > 600 x 109/L
   * Alanine-Aminotransferase (ALT) or Aspartate-Aminotransferase (AST) > 2x upper limit normal
   * Alkaline Phosphatase > 2x upper limit normal
   * Serum Creatinine > upper limit normal
6. History of gastrointestinal surgery, with the exception of appendectomy unless it was performed within the previous 12 months.
7. History of cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome (within the previous 12 months).
8. History of adverse reaction or allergy to Mesalazine or other salicylates.
9. Acute diarrhoea or constipation in the 14 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion is to be determined on the first study day. Diarrhoea will be defined as the passage of liquid faeces and/or qa stool frequency of > 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
10. Donation of blood within the previous three months.
11. Positive HBV-Antigen (Hepatitis-B), HCV-Antibody (Hepatitis-C) or HIV-Antibody (Human Immunodeficiency Virus) results.
12. Over-the-counter (OTC) and prescription medication (including laxatives, vitamin-pills and natural herbal remedies) between screening visit (visit 1) and completion of the study. Occasional paracetamol or acetyl-salicyl-acid is permitted.
13. Failure to satisfy the Principle Investigator to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Tablet release | 3 days

SECONDARY OUTCOMES:
Maximal Plasma Concentration (Cmax) | 3 days
Time to reach Cmax (Tmax) | 3 days
Area under the concentration-time curve | 3 days
Elimination rate constant (k) | 3 days
Lag time (t-lag) | 3 days